CLINICAL TRIAL: NCT00299143
Title: Pilot Study on Shear-induced Platelet Aggregation in Acute Coronary Syndromes
Acronym: REACS
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Principal Investigator, Nadine Ajzenberg, professor, Institut National de la Santé Et de la Recherche Médicale, France
Other Study IDs: RBM 04-24
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Angina, Unstable
Keywords: SIPA; acute coronary syndrome
MeSH Terms: conditions — Angina, Unstable; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, plasma, urines
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether shear-induced platelet aggregation is able to discriminate first acute coronary syndrome (ACS) from recurrent ACS

DETAILED DESCRIPTION:
Predictive factors of recurrence of ACS are not well determined. Platelet aggregation and leucocyte activation seem to be involved in the pathogenesis. The aim of our study is to compare SIPA, platelet activation and platelet-leucocytes aggregates on the onset of the ACS and 3 months later in 2 groups of patients scheduled for a first episode of ACS or recurrent ACS .

ELIGIBILITY:
Inclusion Criteria:

over 18 years old. informed consent signed. acute coronary syndrome not associated with co-morbidity as bleeding diathesis or myocardial infarction during the procedure.

clinical symptoms in agreement with myocardial infarction during the preceding 24 hours.

CK OR troponin elevation and one or more of the following criteria: ECG modifications transient ST elevation>1 mm. new inversion of ST <1 mm on 2 contiguous derivations.

Exclusion criteria:

Acute coronary syndrome with persistent ST elevation. Angioplasty in emergency before blood sampling. Inflammatory disease or cancer. Coagulation abnormalities. Antiphospholipid syndrome. Treatment by vitamin K antagonist. Severe disease with life expectancy lower than 2 years. One-year follow up impossible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in the intensive care unit with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2005-06; Primary Completion 2009-09 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Steg, Professor, Study Director — APHP; Nadine Ajzenberg, Dr, Principal Investigator — APHP, INSERM
Locations (1):
- Bichat Hospital, Paris, France